CLINICAL TRIAL: NCT01846260
Title: Predictive Value of the Distress Thermometer as a Predictive Screening Instrument to Detect Cancer-related Cognitive Impairment in Cancer Patients
Acronym: CONCEPT
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Medical Oncologist, General Hospital Groeninge
Other Study IDs: AZGS2013021
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Cancer Patients Eligible for a Treatment With Curative Intent; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Cognitive impairment associated with chemotherapy is an important reported post-treatment side-effect among breast and other cancer survivors. As some patients report cognitive complaints before the administration of their therapy, some authors suggest an association with psychological risk factors such as distress. Distress, a multifactorial unpleasant emotional experience of a psychological (cognitive, behavioral and emotional), social and/or spiritual nature that may interfere with the ability to cope with cancer effectively, its physical symptoms and its treatment, can easily be assessed by the Distress Thermometer.

In this trial we aim to determine if the Distress Thermometer, accompanied by the 38-item Problem List, could predict cancer-related cognitive impairment in patients with hematologic malignancies, and in patients with gynecological, urological, breast, lung or gastro-intestinal cancer receiving curative radiotherapy, chemotherapy, radiochemotherapy, anti-hormonal or targeted therapy.

DETAILED DESCRIPTION:
Design: Prospective, observational study. All cancer patients of the above mentioned cancer types receiving an anticancer treatment with curative intent will be asked to participate to this study. Consenting patients will undergo serial assessment at baseline, and 6 months after inclusion. Patient will be screened by the Distress Thermometer and 38-item Problem List followed by a neuropsychological assessment and self-assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached a minimum age of 18 years at the time of enrolment
* Newly detected histologically confirmed diagnosis of a solid (lung, gastro-intestinal, GIST, urological, prostate, breast, sarcoma or gynecological cancer) or hematologic malignancy
* Patients should receive a treatment with curative intent based on the investigator's judgment or have an expected median overall survival of at least 5 years
* Patients scheduled to receive (adjuvant) radiotherapy, chemotherapy, radiobiotherapy, radiochemotherapy, anti-hormonal or targeted therapy with curative intent
* Patients should be able to adequately communicate in Dutch
* Patients should present with a sufficient mental and physical functional status (according to investigator's judgment and first baseline assessment) for completing the questionnaires and neuropsychological assessment

Exclusion Criteria:

* Patients younger than 18 at the time of enrollment
* Patients who present with a cognitive impairment
* Patient receiving a treatment with palliative intent
* Patients who had surgery in the three weeks preceding the baseline assessment
* Patients diagnosed with primary or secondary brain tumors
* Patients with a prior history of cancer during the last 5 years, with or without chemotherapy or radiotherapy
* Patients suffering from organic brain disease
* Patients with an untreated or unstable major medical condition
* Patients who are alcohol or drug dependent
* Patients showing signs of mental deterioration
* Patients with dementia (DSM-IV criteria)
* Patients with a major psychiatric or neurologic disorder that could potentially invalidate assessment; a prior or current diagnosis of a depressive or anxiety disorder is allowed
* Patients presenting with a condition other than cancer in which fatigue is a prominent symptom (such as chronic fatigue symptom)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of newly diagnosed cancer patients of all ages (≥18 years), presenting with a solid tumour (lung, gastro-intestinal, GIST, urological, prostate, breast, sarcoma or gynecological cancer) or hematologic malignancy, in an early or advanced stage, eligible for systemic treatment (radiotherapy, chemotherapy, radiochemotherapy, radiobiotherapy, anti-hormonal or targeted therapy) with curative intent.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Validation of the Distress Thermometer, accompanied by the 38-item Problem List, as a screening tool to predict cancer-related cognitive impairment, measured through standard neuropsychological testing | 6 months
  The primary objective of this observational study is to validate the Distress Thermometer, accompanied by the 38-item Problem List, as a screening tool to predict cancer-related cognitive impairment, measured through standard neuropsychological testing in cancer patients receiving curative (adjuvant) radiotherapy, chemotherapy, radiochemotherapy, radiobiotherapy, or targeted therapy.

SECONDARY OUTCOMES:
Prevalence of cognitive impairments and distress in all cancer patients included in this study and per cohort in a general hospital in Belgium by use of the Distress Thermometer and neuropsychological assessment | 6 months
Comparison of subjective patient reported symptoms through self-reported measurements with objective neurocognitive test results and to examine the feasibility of these self-report assessment | 6 months
Evaluation of the performance of the distress thermometer to detect cancer-related cognitive impairments over time | 6 months
Determination of a cut-off score for the Distress Thermometer as a screening tool to detect cancer-related cognitive impairments over time by use of Receiver Operating Characteristics (ROC) curve | 6 months
Evaluation of distress scores compared to patients' quality of life post-treatment by use of EORTC QLQ C-30 | 2 years

OTHER OUTCOMES:
Evaluation of lipid profiles at baseline to establish if fatty acid deficiency is associated with chemobrain through analysis of RBC fatty acid composition | 6 months
Evaluation of CRP-levels as a biomarker to predict cancer-related cognitive decline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD, PhD, Principal Investigator — General Hospital Groeninge
Locations (1):
- General Hospital Groeninge, Kortrijk, Belgium

REFERENCES:
- [Result] Lycke M, Pottel L, Pottel H, Ketelaars L, Stellamans K, Van Eygen K, Vergauwe P, Werbrouck P, Goethals L, Schofield P, Boterberg T, Debruyne PR. Predictors of baseline cancer-related cognitive impairment in cancer patients scheduled for a curative treatment. Psychooncology. 2017 May;26(5):632-639. doi: 10.1002/pon.4200. Epub 2016 Aug 1. PMID 27338029
- [Result] Lycke M, Lefebvre T, Pottel L, Pottel H, Ketelaars L, Stellamans K, Eygen KV, Vergauwe P, Werbrouck P, Goethals L, Schofield P, Boterberg T, Debruyne PR. The distress thermometer predicts subjective, but not objective, cognitive complaints six months after treatment initiation in cancer patients. J Psychosoc Oncol. 2017 Nov-Dec;35(6):741-757. doi: 10.1080/07347332.2017.1365798. Epub 2017 Aug 17. PMID 28816636